CLINICAL TRIAL: NCT07098988
Title: A Ph2, Randomized, Blinded, Placebo-Controlled Trial Investigating the Efficacy and Safety of Visugromab Versus Placebo, in Combination With Pembrolizumab, Pemetrexed, and Carboplatin, in 1L Treatment of Participants With Metastatic NSCLC (GDFATHER-NSCLC-01)
Brief Title: Trial Investigating Visugromab in Combination With Immunochemotherapy in 1L Treatment of Participants With Metastatic NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CatalYm GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTL-002-003; 2024-516792-32-01 (EU CTIS Number)
Record Dates: First submitted 2025-07-10; First posted 2025-08-01 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Non-Squamous Non-Small Cell Lung Cancer; Adult Solid Tumor
Keywords: CTL-002; Visugromab; GDF-15
MeSH Terms: interventions — pembrolizumab; Pemetrexed

STUDY DESIGN:
Intervention Model Description: Part A: Safety Run-In Part B and Part C: Randomized Part The randomized part consists of two arms: Visugromab + ICT (Arm A) and Placebo + ICT (Arm B) Participants will be allocated in 2:1 ratio to treatment arm A or B.
Who Masked: Participant, Investigator
Masking Description: Participants, Investigator and Site trial team, Sponsor and Service Providers' trial teams (including Imaging vendor) are blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Visugromab (CTL-002) + Immunochemotherapy Combination (SoC treatment) - Arm A (Experimental): Participants receive Visugromab (recommended dose), Pembrolizumab (200 mg), Pemetrexed (500 mg/m2) intravenous (IV) on Day 1 of every 21-day cycle (every 3 weeks, or Q3W) for up to 35 treatments and Carboplatin target dose Area Under Curve (AUC) 5 (max. dose 750 mg) IV on Day 1 of every 21-day cycle (every 3 weeks, or Q3W) for four cycles.
  Interventions: Biological: Visugromab; Biological: Pembrolizumab 200 mg Q3W; Drug: Pemetrexed 500 mg/m^2; Drug: Carboplatin AUC 5
- Placebo + Immunochemotherapy Combination (SoC treatment) - Arm B (Active Comparator): Participants receive matching placebo for visugromab, Pembrolizumab (200 mg), Pemetrexed (500 mg/m2) intravenous (IV) on Day 1 of every 21-day cycle (every 3 weeks, or Q3W) for up to 35 treatments and Carboplatin target dose Area Under Curve (AUC) 5 (max. dose 750 mg) IV on Day 1 of every 21-day cycle (every 3 weeks, or Q3W) for four cycles.
  Interventions: Drug: Matching placebo for visugromab; Biological: Pembrolizumab 200 mg Q3W; Drug: Pemetrexed 500 mg/m^2; Drug: Carboplatin AUC 5

INTERVENTIONS:
Biological: Visugromab — Participants receive Visugromab (recommended dose) intravenous (IV) on Day 1 of every 21-day cycle (every 3 weeks, or Q3W) for up to 35 treatments.
  Other Names: CTL-002
  Arms: Visugromab (CTL-002) + Immunochemotherapy Combination (SoC treatment) - Arm A
Drug: Matching placebo for visugromab — Participants receive Matching Placebo intravenous (IV) on Day 1 of every 21-day cycle (every 3 weeks, or Q3W) for up to 35 treatments.
  Arms: Placebo + Immunochemotherapy Combination (SoC treatment) - Arm B
Biological: Pembrolizumab 200 mg Q3W — Participants receive Pembrolizumab 200 mg intravenous (IV) on Day 1 of every 21-day cycle (every 3 weeks, or Q3W) for up to 35 treatments after visugromab infusion.
  Other Names: Keytruda®
Drug: Pemetrexed 500 mg/m^2 — Participants receive Pemetrexed 500 mg/m^2 IV on Day 1 of every 21-day cycle (every 3 weeks, or Q3W) for up to 35 treatments.
Drug: Carboplatin AUC 5 — Participants receive Carboplatin target dose Area Under Curve (AUC) 5 (maximum dose 750 mg) on Day 1 of each 21-day cycle for four cycles.

SUMMARY:
This is an exploratory, signal finding, randomized, placebo-controlled, blinded, multi-center Phase 2b trial of the anti GDF-15 antibody Visugromab (CTL-002) versus Placebo, combined with Immunochemotherapy (ICT: Pembrolizumab, Pemetrexed, Carboplatin) in the first-line treatment of participants with newly diagnosed metastatic non-squamous NSCLC. The trial consists of 3 Parts, a non-randomized Safety-run-in part (Part A) and the subsequent randomized Ph2b trial with 2 treatment arms. After the treatment of 15 participants with visugromab at the expansion dose, an interim safety and preliminary efficacy analysis will be conducted (Part B), followed by the treatment of the remaining participants (Part C).

ELIGIBILITY:
Main Inclusion Criteria:

* Histologically confirmed, newly diagnosed stage IV non-squamous NSCLC.
* Demonstrated absence of actionable mutations (e.g., EGFR, ALK, among others) that suggest/require treatment with available targeted agent.
* Measurable disease determined by the local site Investigator/radiology by their assessment per RECIST v1.1.
* Have not received prior systemic treatment for advanced/metastatic NSCLC. Participants who received adjuvant or neoadjuvant therapy are eligible if the adjuvant/neoadjuvant therapy was completed at least 12 months prior to the development of metastatic disease and did not contain any PD 1/PD L1 directed CPI therapy.
* Availability of locally determined PD L1 TPS, determined with a test validated for this purpose, from a biopsy obtained after any potential prior systemic treatment for this disease. Participants with PD-L1 TPS ≥ 50% can only be enrolled in case CPI monotherapy is not clinically indicated.
* Availability of a tissue/histological biopsy for translational research investigations and Informed Consent Form (ICF) for biopsy release for translational research signed by participant. The biopsy has to be obtained after any potential prior systemic treatment for this disease and be available for shipment. A cytological sample is not accepted.
* Age ≥ 18 years on the day of signing the informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Adequate organ function (bone marrow, hepatic, renal function and coagulation).

Main Exclusion Criteria:

* Presence of predominantly squamous cell histology or predominantly neuroendocrine histology NSCLC (mixed tumors will be categorized by the predominant cell type) or presence of small cell lung cancer elements (ineligibility independent of percentage).
* Any acute or chronic major tissue injury that may require maintained GDF 15 function for tissue protection as per Investigator assessment (diagnosed with myocardial infarction, or liver, kidney or other major organ failure, all within < 3 months prior to planned treatment start).
* Major surgery (defined as a surgery which requires general anesthetic and/or involves opening of body cavities), within 4 weeks of the first dose of study drug.
* Received potentially curative radiation therapy to the lung that is > 30 Gy within 6 months prior to the first dose of study drug.
* Received or completed any focal radiotherapy for symptoms within 28 days of the first dose of study drug.
* Expected to require any other form of antineoplastic therapy while on trial.
* Clinically active inflammatory bowel disease, active diverticulitis, intra-abdominal abscess, and/or gastrointestinal obstruction.
* Known history of prior malignancy with the exception that the participant has undergone potentially curative therapy with no evidence of that disease recurrence for 5 years since initiation of that therapy.
* Known or detected clinically active central nervous system (CNS) involvement by NSCLC or other tumors, e.g., with symptomatic metastases and/or carcinomatous meningitis. Participants with CNS involvement may be enrolled with mandatory regular imaging of the brain under protocol-defined conditions.
* Have one of the following cardiovascular risk factors: myocardial infarction in the past 3 months before planned treatment start; uncontrolled heart failure; uncontrolled ventricular arrhythmia; QT interval corrected for heart rate using Fridericia's formula interval ≥ 470 ms regardless of sex; peri/myocarditis in the past 3 months before planned treatment start; history of ischemic stroke in the past 3 months before planned treatment start.
* Any active autoimmune that has required systemic treatment in the past 3 months before planned treatment start (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs).
* Comedication with metformin in participants with type II diabetes.
* Has interstitial lung disease or a history of non-infectious pneumonitis that required systemic steroids or current pneumonitis.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2031-03-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | up to 24 months
  Percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 as assessed by the Investigator at any time during the core trial period

SECONDARY OUTCOMES:
Adverse Events | up to 27 months
  Incidence, type and severity of adverse events, treatment emergent adverse events, treatment-related adverse events and serious adverse events
CR rate | up to 24 months
  Complete response rate
PR rate | up to 24 months
  Partial response rate
DOR | up to 24 months
  Duration of response
ORR | up to 24 months
  Objective response rate
TTR | up to 24 months
  Time-to-response rate
PFS | up to 48 months
  Progression-free survival
OS | up to 48 months
  Overall survival
Participant weight course over time | up to 48 months
Maximum Concentration (Cmax) of visugromab | At designated time points (up to 24 months)
  Cmax is the maximum observed serum concentration of visugromab
Minimum Concentration (Cmin) of visugromab | At designated time points (up to 24 months)
  Cmin is the minimum observed serum concentration of visugromab
Participants' subjective well-being as assessed by Non-Small Cell Lung Cancer Symptom Assessment Questionnaire (NSCLC-SAQ) | up to 27 months
  NSCLC-SAQ is a participant reported outcome with seven (7) items assessing five (5) symptom domains of NSCLC: cough, fatigue, pain, dyspnea, and appetite. Each item is scored individually from 0 ("None/Never") to 4 ("Severe/Always"). The total score is calculated by summing domain scores, which are derived as follows: single-item domains (cough, dyspnea, appetite) use the item score; fatigue uses the mean of two items (or one if only one is answered); pain uses the highest score of two items (or one if only one is answered). The total score ranges from 0-20, with higher scores indicating more severe symptoms. If any domain score is missing, a total score is not computed.
Participants' quality of life as assessed by 5-day Functional Living Index-Emesis (5-day FLIE) | At designated time points (up to 3 months)
  FLIE consists of 18 items, with 9 items on nausea and 9 items on vomiting. The impact of nausea and vomiting is assessed through their effects on physical and social activities, and emotional well-being. Each item is rated using a visual analog scale (VAS) from 1 to 7 (In some questions, "1" means that nausea or vomiting does not affect the daily life at all, while in other questions, "1" means it affects the daily life a lot). Scoring is calculated per the FLIE Scoring and Administration Manual. Higher scores indicate less impact of nausea and vomiting on daily life. At least 12 of 18 items must be completed to compute the total score.

CONTACTS AND LOCATIONS:
Overall Officials: Felix Lichtenegger, MD, Study Director — CatalYm GmbH
Locations (13):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Yale Cancer Center, New Haven, Connecticut
  - Duke University Medical Center, Durham, North Carolina
- Germany (3):
  - Evangelical Hospital Bethel, Clinic for Internal Medicine, Hematology/Oncology, Palliative Medicine Johannesstift, Bielefeld, North Rhine-Westphalia
  - Clinics Essen-Mitte, Essen, North Rhine-Westphalia
  - Großhansdorf Hospital - Clinical Center for Pulmonology and Thoracic Surgery, Department of Thoracic Oncology, Großhansdorf, Schleswig-Holstein
- Spain (3):
  - University Hospital of Jaen, Jaén, Andalusia
  - Regional University Hospital of Malaga, Málaga, Andalusia
  - University Hospital Lucus Augusti (HULA), Lugo
- Switzerland (3):
  - University Hospital Basel, Basel, Basel
  - Fribourg Cantonal Hospital, Fribourg, Canton of Fribourg
  - Cantonal Hospital Saint Gallen, Clinic of Oncology and Hematology, Sankt Gallen, Canton of St. Gallen

IPD SHARING:
Plan to Share IPD: No